CLINICAL TRIAL: NCT05140161
Title: Hemostasis Assesment After Application of Lyophilisate Collagen in Nail Surgery: a Randomized Controlled Trial
Brief Title: Hemostasis Assesment After Application of Lyophilisate Collagen in Nail Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Antonio Córdoba-Fernández PhD, PhD, Principal Investigator, Clinical Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1206-N-15
Record Dates: First submitted 2021-10-17; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Nails, Ingrown; Coagulation Defect; Bleeding
Keywords: collagen; nail; ingrown; bleeding; surgery
MeSH Terms: conditions — Nails, Ingrown; Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Collagen 1 (Experimental): Medium porosity collagen sponge is used in the operated nail grooves. The hallux is covered with a non-stick dressing, five gauze surrounding it and a cohesive bandage
  Interventions: Device: collagen
- Collagen 2 (Experimental): High porosity collagen sponge is used in the operated nail grooves. The hallux is covered with a non-stick dressing, five gauze surrounding it and a cohesive bandage
  Interventions: Device: collagen
- Control group (No Intervention): No hemostatic device is used in the nail grooves. No hemostatic device is used in the nail grooves. Only non-stick dressing, five gauze pads and cohesive bandage are used

INTERVENTIONS:
Device: collagen — use of hemostatic device in order to reduce bleeding in nail surgery
  Arms: Collagen 1; Collagen 2

SUMMARY:
The objective of this study is to evaluate the hemostatic capacity of two types of collagen hemostatic sponges in nail surgery.

It is a randomized triple-blind clinical trial with two experimental groups (medium porosity collagen and high porosity collagen) and control group ( non collagen).

DETAILED DESCRIPTION:
To evaluate bleeding, all patients with onychocryptosis will be operated on with the same technique.

In the experimental groups, once the surgical procedure has been completed on both edges of the nail, hemostatic collagen will be applied in the experimental groups (experimental group 1- medium porosity collagen and experimental group 2-high porosity collagen) In all groups, including the control, once the intervention was finished, the same bandage was performed with the same number of gauze pads.

At 72 hours, the gauze set will be removed to weigh it using a precision balance and quantitatively evaluate the amount of bleeding.

In this way, a comparative study can be carried out between the 3 groups and determine if there are statistically significant differences or not, and can determine if lyophilized hemostatic collagen is useful in nail surgery and if there are significant differences between both experimental groups, determining if the percentage of porosity in a hemostatic is relevant in the hemostatic effect.

ELIGIBILITY:
Inclusion Criteria:

* STADIUM I, II, or III (Kline classification) without infective onychocryptosis (cellulitis) on both edges of the Hallux
* Susceptible to phenol-alcohol technique with Suppan I modification

Exclusion Criteria:

* Platelet Antiplatelet Therapy
* Oral Anticoagulant Therapy
* History of congenital or acquired Hemorrhagic Syndrome
* Alteration in the following parameters (platelet count, prothrombin time, activated thromboplastin time, and plasma fibrinogen)

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-12-20 (Estimated); Primary Completion 2021-12-29 (Estimated); Study Completion 2022-02-21 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 72 hours after surgery
  The polypropylene non-stick dressing together with 5 gauze pads from the same manufacturer will be weighed using a precision scale. 72 hours after surgery once the cohesive bandage has been removed, the gauze and the non-stick dressing in contact with the wounds will be weighed equally.

SECONDARY OUTCOMES:
Postoperative pain | 72 hours after surgery
  To measure the postoperative pain, an analog chromatic visual scale for self-evaluation of pain (scale from 0 =absence of pain to 10 =unbearable pain) will be used
Postoperative inflammation | 72 hours after surgery
  The digital circumference (in millimeters) will be measured using a flexible millimeter ruler at the level of the proximal nail fold

OTHER OUTCOMES:
Recovery time | 3 weeks after surgery
  Recovery time clinical indicators will be considered when there is absence of drainage, when granulation tissue is covered by a scab, when there were no signs of erythematous tissue without evidence of infection

IPD SHARING:
Plan to Share IPD: No
participant data will only be available to the principal researcher